CLINICAL TRIAL: NCT02456571
Title: Defining the Relevant Immune Checkpoints Expressed on Metastatic Prostate Cancer Circulating Tumor Cells
Brief Title: CTC Immune Checkpoint
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00063296
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group A: men with mCRPC starting sipuleucel-T (Provenge) with or without abiraterone acetate or enzalutamide will have CTC enumeration and immune checkpoint characterization at baseline, 3 months, 4-12 weeks after completion of sipuleucel-T, and at progression.
  Interventions: Device: CTC biomarker expression prevalence
- Group B: men with mCRPC with visceral or high risk disease pre-abiraterone/enzalutamide will have CTC enumeration and immune checkpoint characterization at baseline, 3 months, and progression.
  Interventions: Device: CTC biomarker expression prevalence
- Group C: men with high volume metastatic castration sensitive prostate cancer (mCSPC) starting hormonal therapy and docetaxel chemotherapy or who decline docetaxel chemotherapy will have CTC enumeration and immune checkpoint characterization at baseline, 3 months, and progression.
  Interventions: Device: CTC biomarker expression prevalence
- Group D: men with enzalutamide or abiraterone acetate resistant mCRPC will have CTC enumeration and immune checkpoint characterization at baseline (i.e. progression on enzalutamide or abiraterone acetate) and 4-12 weeks after completion of next therapy (ex. radium-223 or chemotherapy)
  Interventions: Device: CTC biomarker expression prevalence

INTERVENTIONS:
Device: CTC biomarker expression prevalence

SUMMARY:
This pilot study will explore the prevalence of expression of four immune checkpoint biomarkers on circulating tumor cells (CTCs) from men with metastatic prostate cancer that are captured by EpCAM via the CellSearch method, and specifically defined as co expressing DAPI and cytokeratin, and lacking CD45 expression.

ELIGIBILITY:
Patients will be eligible for inclusion in this study only if all of the following criteria apply:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate. Small cell or neuroendocrine tumors of the prostate are also permitted.
2. Clinical or radiographic evidence of progressive metastatic disease, with progression defined as a rising PSA, new metastatic lesions (bone or soft tissue), or radiographic evidence of tumor growth on CT or MRI.
3. Age ≥ 18 years.
4. Ability to understand and the willingness to sign a written informed consent document.

In addition to meeting all of the above criteria, patients must meet all of the criteria for one of the following groups:

A) mCRPC starting sipuleucel-T (Provenge) with or without abiraterone acetate or enzalutamide

1. For patients with adenocarcinoma of the prostate (not applicable for patients with small cell or neuroendocrine tumors of the prostate, or those receiving ADT therapy): Castrate levels of testosterone (≤ 50 ng/dl)
2. Patient planning to start sipuleucel-T.
3. Enrollment prior to the initiation of sipuleucel-T.

B) mCRPC with visceral or high risk disease pre-abiraterone/enzalutamide

1. For patients with adenocarcinoma of the prostate (not applicable for patients with small cell or neuroendocrine tumors of the prostate, or those receiving ADT therapy): Castrate levels of testosterone (≤ 50 ng/dl)
2. Visceral OR high risk disease - must meet one of the following categories:

   * Visceral disease: Radiographic evidence of liver, adrenal, pulmonary, or brain metastases
   * High risk disease: Presence of at least 2 of the following factors:

     * Bone pain requiring opioids
     * Anemia (Hgb <13 g/dL)
     * Bone scan progression at baseline
     * >2 sites of metastatic disease
     * Karnofsky Performance Status (KPS) ≤ 70
     * PSA doubling time <3 months
3. Patient planning to start abiraterone acetate or enzalutamide.
4. Enrollment prior to the initiation of abiraterone acetate or enzalutamide.

C) Newly diagnosed metastatic castration sensitive prostate cancer (mCSPC) starting androgen deprivation therapy

1. Evidence of metastatic disease on radiographic imaging
2. Enrollment within 2 weeks of initiation of androgen deprivation therapy (ADT).
3. Lack of history of hypogonadism

D) Enzalutamide or abiraterone acetate resistant mCRPC

1. For patients with adenocarcinoma of the prostate (not applicable for patients with small cell or neuroendocrine tumors of the prostate, or those receiving ADT therapy): Castrate levels of testosterone (≤ 50 ng/dl)
2. Evidence of disease progression on or following enzalutamide or abiraterone acetate, as defined by one of the following:

   * Radiographic evidence of disease progression as defined by new bone scan lesions or growth of existing soft tissue/visceral/lymph node/bone metastases as determined by the investigator
   * Clinical progression of disease with cutaneous lesions or palpable lesions in absence of radiographic progression

Exclusion Criteria:

1. History of intercurrent or past medical or psychiatric illness that would make participation in a blood drawing protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s).
2. Treatment with an anthracycline (including mitoxantrone) within 1 week of CTC collection, as anthracyclines cause auto-fluorescence of cells.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Duke Cancer Institute Patients
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Change in expression of four immune checkpoint biomarkers (PD-L1, PD-L2, B7-H3, and CTLA-4) on circulating tumor cells (CTCs). | Baseline to 12 weeks
Change in expression of four immune checkpoint biomarkers (PD-L1, PD-L2, B7-H3, and CTLA-4) on circulating tumor cells (CTCs). | Baseline to 14 months (expected time of progression)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States